CLINICAL TRIAL: NCT02861924
Title: Réponse à l'Application d'Une Pression Locale en Laser Speckle Imaging Locally Applied Pressure-induced Vasodilatation
Brief Title: Locally Applied Pressure-induced Vasodilatation
Acronym: LAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-A00609-42
Record Dates: First submitted 2016-07-19; First posted 2016-08-10 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- microcirculatory responses (Experimental): Measure microcirculatory responses after localized ischemia obtained by local application of pressure (laser speckle).
  A pressure is applied to the subject's arm. this causes a localized ischemia. the measures responses to this ischemia will be made by the imager speckle (LSCI) give the microvascular perfusion data.
  Interventions: Other: microcirculatory responses

INTERVENTIONS:
Other: microcirculatory responses — The effect of the duration and intensity of the pressure; reproducibility and correlation with ischemic hyperemia post.
  measurements are made with the Imager SPECKLE imager (LSCI) give the microvascular perfusion data in arbitrary units called perfusion units (UP).

SUMMARY:
Measure microcirculatory responses after localized ischemia obtained by local application of pressure (laser speckle).

DETAILED DESCRIPTION:
Measure microcirculatory responses after localized ischemia obtained by local application of pressure (laser speckle). The purpose of this study is to perform measurements of the methodological points made.

The study will investigate :

* The effect of the duration and intensity of the pressure
* The reproducibility of measurements
* The correlation with ischemic hyperemia post

ELIGIBILITY:
Inclusion Criteria:

* subjects without vascular pathology

Exclusion Criteria:

* pregnancy
* allergy tape

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
microcirculatory response to local pressure. Measurements are made with the Imager SPECKLE imager (LSCI) give the microvascular perfusion data in arbitrary units called perfusion units (UP). | 2 hours
  Measurements are made with the Imager SPECKLE imager (LSCI) give the microvascular perfusion data in arbitrary units called perfusion units (UP).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ABRAHAM, professor, Principal Investigator — UH ANGERS
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henni S, Hersant J, Loufrani L, Duval G, Humeau-Heurtier A; SIMS Group; Riou J, Abraham P; SOCOS Group. Painless local pressure application to test microvascular reactivity to ischemia. Microvasc Res. 2019 Mar;122:13-21. doi: 10.1016/j.mvr.2018.10.013. Epub 2018 Nov 3. PMID 30399363